CLINICAL TRIAL: NCT04610229
Title: Safety of Intensity-modulated Radiotherapy Treatment With Inhomogeneous Dose Distribution in Patients With Relapsed High-grade Gliomas.
Brief Title: Safety of IMRT Treatment With Inhomogeneous Dose in Patients With Relapsed High-grade Gliomas.
Acronym: GLIORAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GLIORAD_15-18
Record Dates: First submitted 2020-08-25; First posted 2020-10-30 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2019-04

CONDITIONS: Glioblastoma Multiforme; Glioblastoma; Glioblastoma, Adult
Keywords: dose painting; hypofractionation; recurrent glioblastoma; tumour; radiotherapy; retreatment; brain
MeSH Terms: conditions — Glioblastoma; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treated with hypofractionation (Experimental): 1
  Interventions: Radiation: Hypofractionation guioded by dose painting

INTERVENTIONS:
Radiation: Hypofractionation guioded by dose painting — 1

SUMMARY:
Relapsed GBMs have a life expectancy of a few months and re-radiation has proven to be safe in terms of toxicity and effective in increasing OS. One of our studies [Ciammella P, 2013, 8:222] reported a median survival of 9.5 months in patients with recurrent GBM and treated with stereotactic radiotherapy with a total dose of 25 Gy in 5 consecutive sessions, in which the dose was prescribed to 70% isodose with a homogeneous gradient towards the center of the target volume. The identification with functional imaging of specific areas with higher tumor cell density, and the possibility of delivering precisely, thanks to the most advanced therapy units, different doses to the different sub-volumes, can lead to an increase in the maximum dose that can be delivered at the expense of the most aggressive areas (with a greater effect on the tumor), compared to smaller doses in areas with lower signal alteration. This selectivity of the doses should allow an increase in the efficacy of the therapy and therefore a hypothetical increase in local control, compared to a radio-induced toxicity on the surrounding healthy tissues almost comparable to that achieved with the previous hypofractionated treatments [Ciammella P, 2013]. In fact, delivering many high doses to the entire volume would result in an excess of radio-induced necrosis within the irradiated regions with high dose, as well as the impossibility of minimizing the doses on healthy areas and / or on non-neoplastic critical areas keeping them at internal dose ranges related to minimal and acceptable toxicity levels. Since there are no studies providing clear indications on the acute and late toxicity of irradiated healthy tissues that have already been the subject of a first course of radiotherapy (STUPP), the choice of safety is the primary objective of the study.

DETAILED DESCRIPTION:
It is an exploratory, prospective, experimental, monocentric study. Having identified a main safety endpoint (toxicity of radiotherapy treatment) and in the absence of data currently available from previous studies and useful for sizing the sample, the sample is defined according to opportunity and feasibility criteria, (12 cases), with a drawing (3 cases + 3 cases + 6 cases) which provides for two intermediate safety assessment steps one month after the end of the third and sixth patient treatment. The study will be continued only in case of positive evaluation of both steps. For each individual patient the treatment is considered completed if: a) the experimental radiotherapy treatment has been completed; b) the first follow-up radiological assessment (NMR) was performed; c) the study treatment was prematurely interrupted due to lack of efficacy (documented disease progression) or unacceptable toxicity.

* Treatment: the treatment foreseen by the protocol foresees the planning and the execution of a hypofractionated radiotherapy (RT) treatment, administered in 5 daily sessions, with intensity modulated technique and inhomogeneous distribution of the dose guided by the diffusion images obtained with magnetic resonance (RM). The radiotherapy treatment must start within 7 days from the date of execution of the centering MRI which will include both the classic morphological sequences with administration of contrast medium and functional ones. In selected cases and according to clinical judgment it will be possible to request the revision of the anatomopathological and radiological findings.
* Radiation technique: for each patient, a radiotherapy treatment plan will be performed with conformed techniques such as intensity-modulated radiotherapy (IMRT) with dose redistribution: dose-painting.
* Positioning and immobilization of the patient: the patient must be treated in a supine position. The arms must be positioned along the body. The use of a knee support is recommended. The garment will be immobilized with a thermoplastic mask and corresponding neck rest supports.
* TC and planning RM: the planning CT should be acquired possibly with reduced layer thickness that contains the entire volume of the skull and the upper part of the shoulders. This is done to allow the possibility of planning non-coplanar type treatments. The last follow-up MRI, or the radiotherapy centering RM, composed of standard and functional sequences, is used for planning, in addition to those that the neuroradiologist will have considered useful to better characterize the clinical case under examination. More details on this are described in the Technical Annex.
* Target volume and organs at risk (OAR): the following target volumes must be identified: • Gross tumor volume (GTV): it is defined using and combining the conventional and advanced sequences of the NMR. • Planning target volume (PTV): it is represented by the GTV with three-dimensional expansion between 0 and 5 mm according to the problems highlighted during the tumor segmentation phase. See the Technical Annex in this regard.
* The following risky organs (OAR) must be identified: • Optical nerves: the definition of the related planning risk volume is also suggested (PRV: organ at risk with three-dimensional expansion; this margin must be chosen taking into account the acquisition thickness of the centering TC and the chosen GTV-PTV expansion margin). • chiasm. We also suggest the definition of the relative PRV (organ at risk with three-dimensional expansion; this margin must be chosen taking into account the acquisition thickness of the centering CT and the chosen GTV-PTV expansion margin). • retinas. We also suggest the definition of the relative PRV (organ at risk with three-dimensional expansion; this margin must be chosen taking into account the acquisition thickness of the centering CT and the chosen GTV-PTV expansion margin). Alternatively the eye globes can be surrounded. • Encefalic trunk.
* The following secondary OARs must be identified: • Lenses / Crystalline. We also suggest the definition of the relative PRV (organ at risk with three-dimensional expansion; this margin must be chosen taking into account the acquisition thickness of the centering CT and the chosen GTV-PTV expansion margin). • Healthy brain tissue. It is represented by the encephalon volume minus the PTV. • Screw. We also suggest the definition of the relative PRV (organ at risk with three-dimensional expansion; this margin must be chosen taking into account the acquisition thickness of the centering CT and the chosen GTV-PTV expansion margin).
* Dose prescription: i) Dose to the target: the prescription dose foresees a minimum dose of 30 Gy (6 Gy per session) for the areas with the highest ADC with a gradual increase in the dose of the lower ADC areas. The maximum hypothesized dose is 50 Gy, with a dose of 10 Gy per session to no more than 1cc of the irradiated brain tissue. The treatment plan, however, will be processed in the following order of priority: 1. Compliance with dose limits for primary OARs. 2. PTV coverage. 3. Compliance with dose limits for secondary OARs.
* Dose limits for primary risk organs: in the scientific literature there are various studies that indicate the dose limits of the organs at risk for brain radiation treatments.

ELIGIBILITY:
Inclusion Criteria:

relapsed GBM after standard surgery-radio-chemotherapy treatment or other therapeutic lines or GBM secondary to anaplastic astrocytomas previously treated with RT and chemotherapy or recurrent anaplastic astrocytomas

* ECOG Performance Status 0-2, Performance Karnofsky Score> 60.
* Written informed consent.
* Life expectancy> 3 months.
* Availability of the patient to be followed for all the phases of the chemotherapy treatment and for the subsequent follow-up.-

Exclusion Criteria:

Patients with KPS <70%.

* Participation in other studies that involve the administration of experimental drugs or explicitly exclude the possibility of participating in other studies in general or in studies whose features include aspects of this study.
* Any concurrent medical or psychological condition that may prevent participation in the study or compromise the ability to provide informed consent.
* Pregnant and lactating patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2019-08-12 (Actual); Study Completion 2019-08-26 (Actual)

PRIMARY OUTCOMES:
Number of adverse events occuring after treatment | 3 months
  Evaluation of side effects in order to assess the risk / benefit ratio. Values greater than G3 according to the CTCAE v.4.0 scale will be considered adverse events.

SECONDARY OUTCOMES:
Local control according to the RANO criteria | 3 months
  Evaluation of the response rate according to the RANO criteria
Incidence of radionecrosis | 3 months
  Incidence of treatment-related radionecrosis measured with advanced magnetic resonance sequences.
Proportion of patients alive 3 months after treatment | 3 months
  Evaluation of survival in retreated patients
Change in health related global quality of life (QOL) | 3 months
  Health related QOL (HRQOL) evaluations using the EORTC QLQ-C30 (version 3) questionnaire. Raw scores will be transformed to a linear scale ranging from 0 to 100 (according to the standard EORTC) with a higher score representing a higher level for functioning or higher livel of symptomatology or problems.
  [N.W.Scott et al, Qual Life, 2009, 18:381-388]
Change in health related quality of life (QOL) for brain cancer disease | 3 months
  Brain cancer specific QOL evaluated by using the EORTC QLQ - BN20 questionnaire. Raw scores will be transformed to a linear scale ranging from 0 to 100 (according to the standard EORTC) with a higher score representing a higher level for functioning or higher livel of symptomatology or problems.
  [MJB Taphoorn et al, EJC, 2010, 46:1033-1040]
Proportion of patients with disease progression 3 months after treatment | 3 months
  Evaluation of disease progression in retreated patients

CONTACTS AND LOCATIONS:
Overall Officials: MAURO MI IORI, PhD, Principal Investigator — MEDICAL PHYSISCS UNIT AUSL IRCCS REGGIO EMILIA ITALY; PATRIZIA PC CIAMMELLA, MD, Study Chair — RADIOTHERAPY UNIT AUSL IRCCS REGGIO EMILIA ITALY
Locations (1):
- Radiotherapy Unit Ausl Irccs Reggio Emilia, Reggio Emilia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ciammella P, Podgornii A, Galeandro M, D'Abbiero N, Pisanello A, Botti A, Cagni E, Iori M, Iotti C. Hypofractionated stereotactic radiation therapy for recurrent glioblastoma: single institutional experience. Radiat Oncol. 2013 Sep 25;8:222. doi: 10.1186/1748-717X-8-222. PMID 24066926
- [Background] Franco P, De Bari B, Ciammella P, Fiorentino A, Chiesa S, Amelio D, Pinzi V, Bonomo P, Vagge S, Fiore M, Comito T, Cecconi A, Mortellaro G, Bruni A, Trovo M, Filippi AR, Greto D, Alongi F; AIRO Giovani Italian Association of Radiation Oncology, Young Members Working Group. The role of stereotactic ablative radiotherapy in oncological and non-oncological clinical settings: highlights from the 7th Meeting of AIRO--Young Members Working Group (AIRO Giovani). Tumori. 2014 Nov-Dec;100(6):e214-9. doi: 10.1700/1778.19280. PMID 25688503
- [Background] Filippi AR, Ciammella P, Piva C, Ragona R, Botto B, Gavarotti P, Merli F, Vitolo U, Iotti C, Ricardi U. Involved-site image-guided intensity modulated versus 3D conformal radiation therapy in early stage supradiaphragmatic Hodgkin lymphoma. Int J Radiat Oncol Biol Phys. 2014 Jun 1;89(2):370-5. doi: 10.1016/j.ijrobp.2014.01.041. Epub 2014 Mar 7. PMID 24613810
- [Background] Navarria P, Minniti G, Clerici E, Tomatis S, Pinzi V, Ciammella P, Galaverni M, Amelio D, Scartoni D, Scoccianti S, Krengli M, Masini L, Draghini L, Maranzano E, Borzillo V, Muto P, Ferrarese F, Fariselli L, Livi L, Pasqualetti F, Fiorentino A, Alongi F, di Monale MB, Magrini S, Scorsetti M. Re-irradiation for recurrent glioma: outcome evaluation, toxicity and prognostic factors assessment. A multicenter study of the Radiation Oncology Italian Association (AIRO). J Neurooncol. 2019 Mar;142(1):59-67. doi: 10.1007/s11060-018-03059-x. Epub 2018 Dec 4. PMID 30515706
- [Background] Ciammella P, Galeandro M, D'Abbiero N, Podgornii A, Pisanello A, Botti A, Cagni E, Iori M, Iotti C. Hypo-fractionated IMRT for patients with newly diagnosed glioblastoma multiforme: a 6 year single institutional experience. Clin Neurol Neurosurg. 2013 Sep;115(9):1609-14. doi: 10.1016/j.clineuro.2013.02.001. Epub 2013 Feb 26. PMID 23453151
- [Background] Orlandi M, Botti A, Sghedoni R, Cagni E, Ciammella P, Iotti C, Iori M. Feasibility of voxel-based Dose Painting for recurrent Glioblastoma guided by ADC values of Diffusion-Weighted MR imaging. Phys Med. 2016 Dec;32(12):1651-1658. doi: 10.1016/j.ejmp.2016.11.106. Epub 2016 Dec 16. PMID 27989415

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-16): https://cdn.clinicaltrials.gov/large-docs/29/NCT04610229/Prot_SAP_000.pdf